CLINICAL TRIAL: NCT02104583
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Dose Ranging, Parallel Group Study to Evaluate the Effect of GS-6615 on Ventricular Arrhythmia in Subjects With Implantable Cardioverter-Defibrillator (ICD) or Cardiac Resynchronization Therapy-Defibrillator (CRT-D)
Brief Title: Evaluating Ventricular Arrhythmia in Subjects With Implantable Cardioverter Defibrillator or Cardiac Resynchronization Therapy-Defibrillator
Acronym: TEMPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-356-0101; 2013-004430-15 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Ventricular Arrhythmia
Keywords: VT; VF; Ventricular Tachycardia; Ventricular Fibrillation; shock; ATP
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Shock | interventions — eleclazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Eleclazine 3 mg (Experimental): Participants will receive a single loading dose of eleclazine 30 mg on Day 1, followed by eleclazine 3 mg daily as maintenance for up to approximately 20 months.
  Interventions: Drug: Eleclazine
- Eleclazine 6 mg (Experimental): Participants will receive a single loading dose of eleclazine 30 mg on Day 1, followed by eleclazine 6 mg daily as maintenance for up to approximately 20 months.
  Interventions: Drug: Eleclazine
- Placebo (Placebo Comparator): Participants will receive a single loading dose of placebo to match eleclazine on Day 1, followed by placebo to match eleclazine once daily for up to approximately 20 months.
  Interventions: Drug: Placebo to match eleclazine

INTERVENTIONS:
Drug: Eleclazine — Eleclazine tablets administered orally
  Other Names: GS-6615
  Arms: Eleclazine 3 mg; Eleclazine 6 mg
Drug: Placebo to match eleclazine — Placebo to match eleclazine tablets administered orally
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of eleclazine (GS-6615) compared to placebo on the overall occurrence of appropriate implantable cardioverter-defibrillator (ICD) interventions (antitachycardia pacing [ATP] or shock) in adults with ICD or cardiac resynchronization therapy-defibrillator (CRT-D).

ELIGIBILITY:
Key Inclusion Criteria:

* Have an ICD or CRT-D implanted for primary or secondary prevention and at least one ICD intervention for ventricular tachycardia/ventricular fibrillation (VT/VF) [shock or ATP] within 60 days prior to screening or a documented VT/VF episode (prior to implantation) within 60 days prior to screening
* Use of highly effective contraception methods if female of childbearing potential or sexually active male
* Must be hemodynamically stable

Key Exclusion Criteria:

* New York Heart Association (NYHA) Class IV heart failure
* Myocardial infarction, unstable angina, coronary artery bypass graft (CABG) surgery or percutaneous coronary intervention (PCI) within 4 weeks prior to screening or during the screening period before randomization
* Hemodynamically significant primary obstructive valvular disease
* History of congenital heart disease
* Inherited arrhythmia such as Brugada syndrome. Individuals with long QT syndrome Type 3 (LQT-3) or hypertrophic cardiomyopathy (HCM) may be considered.
* Individuals who are being considered for cardiac transplantation and are on a cardiac transplant list
* History of seizures or epilepsy
* Cardiac ablation within 3 months prior to screening or planned cardiac ablation during the study
* Severe renal impairment
* Abnormal liver function tests
* Currently taking Class I and Class III antiarrhythmic drugs; such medications should be discontinued 5 half-lives (or 28 days for chronic use of amiodarone) prior to randomization
* Currently taking drugs or products that are strong inhibitors or inducers of CYP3A; such medications should be discontinued 5 half-lives prior to randomization
* Currently taking ranolazine; ranolazine should be discontinued at least 7 days prior to randomization
* Females who are pregnant or are breastfeeding
* Individuals with a subcutaneous ICD
* Body mass index (BMI) ≥ 36 kg/m^2

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (84):
- United States (37):
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Long Beach Memorial Hospital, Long Beach, California
  - Good Samaritan Hospital, Los Angeles, California
  - Radin Cardiovascular Medical Associates, Newport Beach, California
  - Regional Cardiology Associates, Sacramento, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Atlantic Clinical Research Collaborative, Atlantis, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Coastal Cardiology Consultants PA dba Heart and Vascular Institute of Florida, Clearwater, Florida
  - The Heart Institute at Largo, Largo, Florida
  - Charlotte Heart and Vascular Institute, Port Charlotte, Florida
  - Florida Medical Clinic PA, Zephyrhills, Florida
  - Athens Regional Specialty Services, Athens, Georgia
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Mid Michigan Medical Center - Midland, Midland, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Great Falls Clinic, Great Falls, Montana
  - Methodist Physicians Clinic Heart Consultants, Omaha, Nebraska
  - New Mexico Hear Institute, Albuquerque, New Mexico
  - New York Methodist Hospital, Brooklyn, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Ohiohealth Corporation, Columbus, Ohio
  - Capital Area Research, Camp Hill, Pennsylvania
  - CardioVascular Institute, Wormleysburg, Pennsylvania
  - Care New England Health Care, Kent Hospital, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Seton Heart Institute, Austin, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - West Houston Area Clinical Trial Consultants, Houston, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Heart Group Ltd, Falls Church, Virginia
  - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Canada (4):
  - Kingston General Hospital, Kingston, Ontario
  - Chum Hotel Dieu, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke CHUS, Sherbrooke, Quebec
  - QEII Health Sciences Centre, Halifax
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc
  - Charles University Hospital Královské Vinohrady, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, The Heart Center, Copenhagen
  - Gentofte Hospitak, Deparment of Cardiology, Hellerup
  - Odense University Hospital/Department of Cardiology, Odense C
- Germany (6):
  - Vivantes Humboldt Klinikum, Berlin
  - University Medical Center Goettingen, Göttingen
  - University of Heidelberg, Heidelberg
  - Medizinische Klinik und Poliklinik I Abteilung für Kardiologie, Munich
  - Klinikum der Universität Regensburg, Regensburg
  - Gemeinschaftspraxis für Innere Medizin, Riesa
- Hungary (5):
  - State Hospital for Cardiology, Balatonfüred
  - Budai Irgalmasrendi Kórház, Budapest
  - Semmelweis Egyetem, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Zala Megyei Kórház, Zalaegerszeg
- Israel (9):
  - HaEmek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Tel Aviv University/Meir Medical Center, Israel
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (6):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Amphia ziekenhuis, Breda
  - Catharina ziekenhuis, Eindhoven
  - Maastricht University Medical Center, Maastricht
  - St.Antonius Hospital, Nieuwegein
  - Isala, Zwolle
- Poland (11):
  - Samodzielny Publiczny Szpital Kliniczny nr 7 Slaskiego Uniwersytetu Medycznego w Katowicach Górnosla, Katowice
  - Collegium Medicum Uniwersytetu Jagiellonskiego, Krakow
  - Medical University of Lodz, Lodz
  - Mc Tronik Specjalistyczny Gabinet Kontroli Stymulatorow Serca Dr N. Med. Michal Chudzik, Lódz
  - Indywidualna Specjalistyczna Praktyka Lekarska Andrzej Lubinski, Lódz
  - NZOZ Sopockie Centrum badan Kardiolog.ProCordis pawel Miekus, Sopot
  - Indywidualna Specjalistyczna Praktyka Lekarska Jarosław Kaźmierczak, Szczecin
  - Szpital Wolski im Dr Anny Gostynskiej SP ZOZ, Warsaw
  - Warszawski Uniwersytet Medyczny, Warsaw
  - Instytut Kardiologii im Prymasa Tysiaclecia Kardynala Stefana Wyszynskiego, Warsaw
  - Medical University Wroclaw, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Asia. The first participant was screened on 12 September 2014. The last study visit occurred on 14 October 2016.
Pre-assignment Details: 389 participants were screened.
Groups:
- Cohort 1 Eleclazine 3 mg: Participants received single loading dose of eleclazine 30 mg (3 x 10 mg tablets) on Day 1, followed by eleclazine 3 mg tablet once daily as maintenance for up to approximately 22 months.
- Cohort 1 Placebo: Participants received single loading dose of placebo to match eleclazine tablets on Day 1, followed by placebo to match eleclazine tablet once daily for up to approximately 20 months.
- Cohort 2 Eleclazine 3 mg: Participants received single loading dose of eleclazine 30 mg (3 x 10 mg tablets) on Day 1, followed by eleclazine 3 mg tablet once daily as maintenance for up to approximately 14 months.
- Cohort 2 Eleclazine 6 mg: Participants were randomized to receive single loading dose of eleclazine 30 mg (3 x 10 mg tablets) on Day 1, followed by eleclazine 6 mg (2 x 3 mg tablets) once daily as maintenance for up to approximately 14 months.
- Cohort 2 Placebo: Participants received single loading dose of placebo to match eleclazine tablets on Day 1, followed by placebo to match eleclazine tablets once daily for up to approximately 14 months.
Period: Overall Study
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo
Started | 48 | 46 | 70 | 74 | 75
Completed | 30 | 35 | 54 | 57 | 63
Not Completed | 18 | 11 | 16 | 17 | 12
Not completed — New ICD or CRT-D implanted | 2 | 0 | 1 | 0 | 0
Not completed — Death | 2 | 1 | 3 | 3 | 5
Not completed — Subject required cardiac ablation | 6 | 4 | 4 | 5 | 4
Not completed — Subject required prohibited medication | 0 | 1 | 1 | 0 | 1
Not completed — Withdrew Consent | 3 | 2 | 0 | 2 | 1
Not completed — Investigator's Discretion | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 6 | 6 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Randomized but Never Treated | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Analysis set included participants who were randomized into the study.
Groups:
- Cohort 2 Eleclazine 6 mg: Participants received single loading dose of eleclazine 30 mg (3 x 10 mg tablets) on Day 1, followed by eleclazine 6 mg (2 x 3 mg tablets) once daily as maintenance for up to approximately 14 months.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo | Total
Number analyzed (Participants) | 48 | 46 | 70 | 74 | 75 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
  years
    number analyzed (Participants) | 48 | 46 | 70 | 73 | 75 | 312
    (all) | 65 (10.4) | 64 (9.6) | 65 (10.8) | 65 (8.3) | 64 (9.4) | 65 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants in the Safety Analysis Set were analyzed.
  Participants
    number analyzed (Participants) | 48 | 46 | 70 | 73 | 75 | 312
    Female | 4 | 5 | 8 | 7 | 8 | 32
    Male | 44 | 41 | 62 | 66 | 67 | 280
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants in the Safety Analysis Set were analyzed.
  Participants
    Race: number analyzed (Participants) | 48 | 46 | 70 | 73 | 75 | 312
    Race: Black | 1 | 1 | 0 | 2 | 1 | 5
    Race: White | 47 | 45 | 70 | 70 | 71 | 303
    Race: Not permitted | 0 | 0 | 0 | 1 | 2 | 3
    Race: Other | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants in the Safety Analysis Set were analyzed.
  Participants
    Ethnicity: number analyzed (Participants) | 48 | 46 | 70 | 73 | 75 | 312
    Ethnicity: Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 2
    Ethnicity: Not Hispanic or Latino | 47 | 45 | 70 | 71 | 73 | 306
    Ethnicity: Not Permitted | 0 | 1 | 0 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 20 | 24 | 24 | 117
  Poland | 6 | 7 | 18 | 11 | 15 | 57
  Israel | 9 | 8 | 6 | 9 | 6 | 38
  Hungary | 3 | 4 | 9 | 10 | 9 | 35
  Germany | 0 | 1 | 7 | 7 | 9 | 24
  Canada | 0 | 0 | 3 | 3 | 6 | 12
  Netherlands | 0 | 0 | 4 | 5 | 3 | 12
  Denmark | 2 | 0 | 3 | 4 | 1 | 10
  Czechia | 3 | 2 | 0 | 1 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Occurrence (Total Number) of Appropriate Implantable Cardioverter-Defibrillator Device (ICD) Interventions (Anti-Tachycardia Pacing or Shock) Through Week 24
Time Frame: Randomization up to 24 weeks
Population: Participants in the Full Analysis Set-ICD [all participants who were randomized into the study and received at least 1 dose of study medication, restricted to participants who had at least 1 postbaseline ICD/cardiac resynchronization therapy-defibrillator (CRT-D) interrogation] with available data were analyzed.
Measure: Mean (Standard Deviation); unit: events
Groups:
- Cohorts 1 and 2, Eleclazine 3 mg: All randomized participants across cohorts 1 and 2 who received single loading dose of eleclazine 30 mg on Day 1, followed by eleclazine 3 mg daily as maintenance for up to approximately 22 months.
- Cohorts 1 and 2, Placebo: All randomized participants across cohorts 1 and 2 who received single loading dose of placebo to match eleclazine on Day 1, followed by placebo to match eleclazine once daily for up to approximately 20 months.
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo | Cohorts 1 and 2, Eleclazine 3 mg | Cohorts 1 and 2, Placebo
Number analyzed (Participants) | 48 | 46 | 69 | 73 | 75 | 117 | 121
events | 3.3 (6.99) | 1.9 (3.79) | 2.6 (6.8) | 1.1 (2.09) | 1.5 (3.92) | 2.8 (6.86) | 1.7 (3.86)
Statistical Analysis 1: Comparison: Cohorts 1 and 2, Eleclazine 3 mg vs Cohorts 1 and 2, Placebo; The primary analysis of overall occurrence of appropriate ICD interventions through Week 24 was performed using a generalized linear model assuming a negative binomial distribution and log link. This model included terms for treatment, implanted device (ICD or CRT-D) and region [US or rest of world (ROW)]; Test type: Superiority; p = 0.152, generalized linear model; Eleclazine : Placebo Incident Rate Ratio = 1.52, 95% CI 2-sided [0.86 to 2.71]
Statistical Analysis 2: Comparison: Cohort 2 Eleclazine 6 mg vs Cohort 2 Placebo; The primary analysis of overall occurrence of appropriate ICD interventions through Week 24 was performed using a generalized linear model assuming a negative binomial distribution and log link. This model included terms for treatment, implanted device (ICD or CRT-D) and region [US or ROW]; Test type: Superiority; p = 0.662, generalized linear model; Eleclazine : Placebo Incident Rate Ratio = 0.82, 95% CI 2-sided [0.34 to 1.97]
Statistical Analysis 3: Comparison: Cohort 2 Eleclazine 3 mg vs Cohort 2 Placebo; The primary analysis of overall occurrence of appropriate ICD interventions through Week 24 was performed using a generalized linear model assuming a negative binomial distribution and log link. This model included terms for treatment, implanted device (ICD or CRT-D) and region [US or ROW; Test type: Superiority; p = 0.618, generalized linear model; Eleclazine : Placebo Incident Rate Ratio = 1.24, 95% CI 2-sided [0.54 to 2.86]

2. Secondary Outcome: Overall Occurrence (Total Number) of Appropriate ICD Interventions (ATP or Shock) Through End of Study
Time Frame: Randomization up to 22 months
Population: Participants in the Full Analysis Set-ICD with available data were analyzed.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo | Cohorts 1 and 2, Eleclazine 3 mg | Cohorts 1 and 2, Placebo
Number analyzed (Participants) | 48 | 46 | 69 | 73 | 75 | 117 | 121
events | 5.0 (7.92) | 7.2 (20.89) | 3.8 (8.82) | 1.2 (2.11) | 2.0 (5.55) | 4.3 (8.45) | 4.0 (13.75)

3. Secondary Outcome: Change From Baseline in Premature Ventricular Complex (PVC) Count as Assessed by Continuous Electrocardiogram (cECG) Monitoring
Description: PVC count per 48 hours was obtained from cECG readings at Baseline and Week 12. Change in PVC from baseline was measured in units of number of episodes/48 hours. Change from baseline was calculated as the value at Week 12 minus the value at Baseline.
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set (all participants who were randomized into the study and received at least 1 dose of study medication) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: episodes/48 hours
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo
Number analyzed (Participants) | 41 | 40 | 58 | 56 | 63
episodes/48 hours | 4282 (17651.5) | -2347 (8498.8) | -594 (13323.0) | -39 (13575.0) | 1541 (11117.7)

4. Secondary Outcome: Change From Baseline in Nonsustained Ventricular Tachycardia (nsVT) Count as Assessed by Continuous cECG Monitoring
Description: The count of nsVTs per 48 hours was obtained from cECG readings at Baseline and Week 12. Change in nsVT from baseline was measured in units of number of episodes/48 hours. Change from baseline was calculated as the value at Week 12 minus the value at Baseline.
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: episodes/48 hours
Groups:
- Cohort 1 Placebo: Participants received single loading dose of placebo to match eleclazine tabletson Day 1, followed by placebo to match eleclazine tablet once daily for up to approximately 20 months.
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo
Number analyzed (Participants) | 41 | 40 | 58 | 56 | 63
episodes/48 hours | 44 (171.6) | -14 (52.2) | -67 (400.4) | 46 (388.4) | 2 (15.1)

5. Secondary Outcome: Overall Occurrence (Total Number) of Ventricular Tachycardia/Ventricular Fibrillation (VT/VF) (Treated or Untreated) Through Week 24 and End of Study
Time Frame: Randomization up to Week 24; Randomization up to end of study (up to 22 months)
Population: Participants in the Full Analysis Set-ICD with available data were analyzed.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo
Number analyzed (Participants) | 48 | 46 | 69 | 73 | 75
events
  Total Number of Events Through Week 24 | 3.56 (7.554) | 2.07 (3.974) | 2.74 (6.825) | 1.44 (2.779) | 1.61 (3.952)
  Total Number of Events Through End of Study | 5.98 (8.907) | 7.83 (20.949) | 4.07 (9.088) | 1.56 (2.794) | 2.17 (5.574)

6. Secondary Outcome: Overall Occurrence (Total Number) of Electrical Storm Through Week 24 and End of Study
Description: An electrical storm was defined as ≥ 3 separate episodes of ventricular arrhythmia within a 24-hour period terminated by ICD.
Time Frame: Randomization up to Week 24; Randomization up to end of study (up to 22 months)
Population: Participants in the Full Analysis Set-ICD with available data were analyzed.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo
Number analyzed (Participants) | 48 | 46 | 69 | 73 | 75
events
  Total Number of Events Through Week 24 | 0.15 (0.545) | 0.15 (0.631) | 0.23 (0.843) | 0.03 (0.164) | 0.09 (0.408)
  Total Number of Events Through End of Study | 0.21 (0.582) | 0.63 (2.037) | 0.35 (1.041) | 0.03 (0.164) | 0.12 (0.614)

7. Secondary Outcome: Overall Occurrence (Total Number) of Inappropriate ICD Interventions Through Week 24 and End of Study
Time Frame: Randomization up to Week 24; Randomization up to end of study (up to 22 months)
Population: Participants in the Full Analysis Set-ICD with available data were analyzed.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo
Number analyzed (Participants) | 48 | 46 | 69 | 73 | 75
events
  Total Number of Events Through Week 24 | 0.17 (0.753) | 0.15 (0.515) | 0.14 (0.772) | 0.12 (6.22) | 0.39 (2.283)
  Total Number of Events Through End of Study | 0.31 (1.613) | 0.41 (2.072) | 0.16 (0.779) | 0.14 (0.631) | 0.43 (2.395)

8. Secondary Outcome: Change in Left Ventricular Systolic and Diastolic Function as Assessed by Left Ventricular Ejection Fraction (LVEF)
Description: LVEF is a measure of how much blood is pumped out of the left ventricle of the heart. Change from baseline was calculated as the value at Week 12 or 24 minus the value at Baseline.
Time Frame: Baseline to Week 12; Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo
Number analyzed (Participants) | 43 | 45 | 57 | 60 | 66
percentage of blood
  Baseline | 35 (12.8) | 38 (12.4) | 38 (12.1) | 38 (13.3) | 40 (13.5)
  Change at Week 12: number analyzed (Participants) | 41 | 39 | 50 | 46 | 58
  Change at Week 12 | 3 (8.1) | 3 (6.2) | 3 (9.1) | 3 (8.2) | 1 (8.2)
  Change at Week 24: number analyzed (Participants) | 35 | 39 | 44 | 43 | 52
  Change at Week 24 | 1 (12.3) | 2 (8.2) | 3 (10.0) | 1 (10.7) | 0 (8.3)

9. Secondary Outcome: Time From First Dose of Study Drug to the First Occurrence of Appropriate ICD Interventions (ATP or Shock) or Cardiovascular (CV) Death
Description: CV deaths were determined through the adjudication by an external independent clinical event committee (CEC). The deaths that were adjudicated as undetermined were considered cardiovascular related. For each participant, the time from the first dose of study drug to the beginning of the earliest appropriate ICD intervention through the last day on study or, in absence of appropriate ICD interventions, to a CV death was derived as (first event date - first dose date + 1). The participants without appropriate ICD interventions or CV death were censored at the last day on study. As planned, data was reported only for Cohort 2 and combined Cohorts 1 and 2. Time to first occurrence of an appropriate ICD interventions or CV death was analyzed using Kaplan-Meier (KM) estimates.
Time Frame: From first dose of study drug up to 22 months
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo | Cohorts 1 and 2, Eleclazine 3 mg | Cohorts 1 and 2, Placebo
Number analyzed (Participants) | 70 | 73 | 75 | 118 | 121
days | 252.0 [147.0 to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | 243.0 [147.0 to 281.0] | 265.0 [130.0 to 496.0]

10. Secondary Outcome: Time From First Dose of Study Drug to the First Occurrence of CV Hospitalization, Emergency Room (ER) Visit, or CV Death
Description: CV hospitalizations, CV ER visits, and CV deaths were determined through the adjudication by the CEC. The events that were adjudicated as undetermined were considered cardiovascular related. For each participant, the time from the first dose of study drug to the first CV hospitalization or CV ER visit through the last day on study or, in absence of CV hospitalizations or CV ER visits, to a CV death were derived as (first event date - first dose date + 1). The participants without CV hospitalizations, CV ER visits, or CV death were censored at the last day on study. As planned, data was reported only for Cohort 2 and combined Cohorts 1 and 2. Time to first occurrence of CV hospitalization, ER visit, or CV death was analyzed using KM estimates.
Time Frame: From first dose of study drug up to 22 months
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo | Cohorts 1 and 2, Eleclazine 3 mg | Cohorts 1 and 2, Placebo
Number analyzed (Participants) | 70 | 73 | 75 | 118 | 121
days | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored.

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose date (maximum: approximately 96.1 weeks) plus 30 days
Description: Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1 Eleclazine 3 mg | Cohort 1 Placebo | Cohort 2 Eleclazine 3 mg | Cohort 2 Eleclazine 6 mg | Cohort 2 Placebo
Serious Adverse Events (participants affected / at risk) | 27/48 | 25/46 | 28/70 | 26/73 | 26/75
Other Adverse Events (participants affected / at risk) | 32/48 | 26/46 | 42/70 | 34/73 | 33/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Eleclazine 3 mg (N=48) | Cohort 1 Placebo (N=46) | Cohort 2 Eleclazine 3 mg (N=70) | Cohort 2 Eleclazine 6 mg (N=73) | Cohort 2 Placebo (N=75)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Acute right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Anginal equivalent (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 4 | 1 | 4
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 3 | 2
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 0 | 1 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 1 | 1 | 2 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 2 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 3 | 2 | 5 | 2 | 5
Ventricular fibrillation (Cardiac disorders) | 3 | 3 | 0 | 2 | 1
Ventricular flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 11 | 10 | 7 | 10 | 8
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Coeliac artery compression syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 2 | 1
Phantom shocks (General disorders) | 0 | 0 | 0 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Endocarditis pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 3
Septic shock (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Anticoagulation drug level below therapeutic (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Parosmia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 1
Device inappropriate shock delivery (Product Issues) | 0 | 0 | 1 | 0 | 0
Device malfunction (Product Issues) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 3 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Eleclazine 3 mg (N=48) | Cohort 1 Placebo (N=46) | Cohort 2 Eleclazine 3 mg (N=70) | Cohort 2 Eleclazine 6 mg (N=73) | Cohort 2 Placebo (N=75)
Atrial fibrillation (Cardiac disorders) | 4 | 2 | 4 | 2 | 3
Ventricular tachycardia (Cardiac disorders) | 8 | 2 | 8 | 7 | 9
Constipation (Gastrointestinal disorders) | 4 | 1 | 2 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 5 | 4 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 4 | 3 | 2
Asthenia (General disorders) | 3 | 1 | 1 | 3 | 1
Chest discomfort (General disorders) | 4 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 3 | 3 | 4 | 2
Fatigue (General disorders) | 5 | 7 | 6 | 3 | 5
Oedema peripheral (General disorders) | 3 | 3 | 2 | 2 | 3
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 4 | 1 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 5 | 1
Blood magnesium decreased (Investigations) | 3 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 3 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 5 | 4 | 6 | 8 | 2
Headache (Nervous system disorders) | 4 | 2 | 3 | 3 | 3
Syncope (Nervous system disorders) | 2 | 4 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 3 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 5 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 7 | 2 | 5
Hypotension (Vascular disorders) | 3 | 2 | 4 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years